CLINICAL TRIAL: NCT02295553
Title: Co-administration of Ketamine and Propofol for Upper Endoscopy in Children: a Dose-finding Study
Brief Title: Ketamine and Propofol for Upper Endoscopy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Jason Hayes, Staff Anaesthesiologist, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1000036780
Record Dates: First submitted 2013-12-12; First posted 2014-11-20 (Estimated); Results first posted 2019-06-10 (Actual); Last update posted 2019-06-10 (Actual); Status verified 2019-03

CONDITIONS: Anesthesia
Keywords: Ketamine; Propofol; Children; Pediatrics; Upper endoscopy
MeSH Terms: interventions — Ketamine; Propofol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Ketamine 0 mg/kg (Experimental): Ketamine dose will be 0 mg/kg. Propofol dose for the first patient will be 4 mg/kg. Doses for the subsequent patients will increase or decrease by 1.6 mg/kg using the Dixon Up and Down method.
  Interventions: Drug: Propofol
- Ketamine 0.25 mg/kg (Experimental): Ketamine dose will be 0.25 mg/kg. Propofol dose for the first patient will be 3 mg/kg. Doses for the subsequent patients will increase or decrease by 1.2 mg/kg using the Dixon Up and Down method.
  Interventions: Drug: Ketamine; Drug: Propofol
- Ketamine 0.5 mg/kg (Experimental): Ketamine dose will be 0.5 mg/kg. Propofol dose for the first patient will be 2.5 mg/kg. Doses for the subsequent patients will increase or decrease by 0.8 mg/kg using the Dixon Up and Down method.
  Interventions: Drug: Ketamine; Drug: Propofol
- Ketamine 1.0 mg/kg (Experimental): Ketamine dose will be 1.0 mg/kg. Propofol dose for the first patient will be 2 mg/kg. Doses for the subsequent patients will increase or decrease by 0.4 mg/kg using the Dixon Up and Down method.
  Interventions: Drug: Ketamine; Drug: Propofol

INTERVENTIONS:
Drug: Ketamine
  Arms: Ketamine 0.25 mg/kg; Ketamine 0.5 mg/kg; Ketamine 1.0 mg/kg
Drug: Propofol

SUMMARY:
The purpose of this study is to examine the dose-response relationship of ketamine in combination with propofol.

DETAILED DESCRIPTION:
Direct visualization of the esophagus, stomach and small intestine is performed using a scope that is inserted while the patient is under under deep sedation or general anesthesia. The most common method of providing general anesthesia for upper endoscopy is intravenous administration of medications such as propofol, often in combination with other medications such as fentanyl, midazolam, remifentanil or ketamine. One study found that the combination of propofol and ketamine provides better conditions (less patient movement, more stable heart and breathing) but more side effects afterwards compared to propofol and fentanyl.

ELIGIBILITY:
Inclusion Criteria:

* Age 3-13 years
* Receiving general anesthesia for upper endoscopy

Exclusion Criteria:

* Known or possible difficult airway
* BMI > 35
* Weight < 10 kg
* Sedative premedication required
* Known contraindication to ketamine or propofol

Ages: 3 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 56 (Actual)
Dates: Start 2013-07 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason Hayes, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Hayes J, Matava C, Pehora C, El-Beheiry H, Jarvis S, Finkelstein Y. Determination of the median effective dose of propofol in combination with different doses of ketamine during gastro-duodenoscopy in children: a randomised controlled trial. Br J Anaesth. 2018 Aug;121(2):453-461. doi: 10.1016/j.bja.2018.03.037. Epub 2018 Jun 5. PMID 30032885

RESULTS

PARTICIPANT FLOW:
Groups:
- Ketamine 0 mg/kg: Ketamine dose will be 0 mg/kg. Propofol dose for the first patient will be 4 mg/kg. Doses for the subsequent patients will increase or decrease by 1.6 mg/kg using the Dixon Up and Down method.
  Propofol
- Ketamine 0.25 mg/kg: Ketamine dose will be 0.25 mg/kg. Propofol dose for the first patient will be 3 mg/kg. Doses for the subsequent patients will increase or decrease by 1.2 mg/kg using the Dixon Up and Down method.
  Ketamine
  Propofol
- Ketamine 0.5 mg/kg: Ketamine dose will be 0.5 mg/kg. Propofol dose for the first patient will be 2.5 mg/kg. Doses for the subsequent patients will increase or decrease by 0.8 mg/kg using the Dixon Up and Down method.
  Ketamine
  Propofol
- Ketamine 1.0 mg/kg: Ketamine dose will be 1.0 mg/kg. Propofol dose for the first patient will be 2 mg/kg. Doses for the subsequent patients will increase or decrease by 0.4 mg/kg using the Dixon Up and Down method.
  Ketamine
  Propofol
Period: Overall Study
Arm/Group | Ketamine 0 mg/kg | Ketamine 0.25 mg/kg | Ketamine 0.5 mg/kg | Ketamine 1.0 mg/kg
Started | 14 | 14 | 14 | 14
Completed | 14 | 14 | 13 | 13
Not Completed | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ketamine 0 mg/kg | Ketamine 0.25 mg/kg | Ketamine 0.5 mg/kg | Ketamine 1.0 mg/kg | Total
Number analyzed (Participants) | 14 | 14 | 13 | 14 | 55
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.4 (2.8) | 8.9 (2.7) | 8.9 (2.1) | 8.9 (2.5) | 8.8 (2.5)
Sex/Gender, Customized [Count of Participants; unit: Participants] | NA — We did not collect information on this demographic | NA — We did not collect information on this demographic | NA — We did not collect information on this demographic | NA — We did not collect information on this demographic | NA — Total not calculated because data are not available (NA) in one or more arms.
Weight [Mean (Standard Deviation); unit: kg] | 30.1 (12.4) | 28.5 (8.9) | 29.5 (0.9) | 30.0 (10.7) | 29.5 (10.3)

OUTCOME MEASURES:

1. Primary Outcome: Dose of Propofol Required to Prevent Movement (Response) to Insertion of Endoscope Into the Patient's Esophagus
Description: The objective is to determine the effective bolus dose in 50% of subjects (ED50) of propofol in combination with ketamine 0, 0.25, 0.5 and 1 mg/kg that produces an adequate depth of anesthesia to prevent minimal or no movement on endoscope insertion in children
Time Frame: This outcome is measured at the time of insertion of the endoscope into the esophagus.
Population: Dose of propofol required to prevent movement upon insertion of endoscope
Measure: Mean (95% Confidence Interval); unit: mg/kg
Arm/Group | Ketamine 0 mg/kg | Ketamine 0.25 mg/kg | Ketamine 0.5 mg/kg | Ketamine 1.0 mg/kg
Number analyzed (Participants) | 14 | 14 | 13 | 14
mg/kg | 6.1 [4.1 to 8.1] | 4.5 [2.9 to 6] | 4.7 [3.1 to 6.2] | 1.1 [0.5 to 1.8]

2. Secondary Outcome: Duration of Apnea After Propofol Administration
Description: The patient will be observed for apnea after propofol is administered until the endoscopy procedure is complete. Duration of apnea will be recorded.
Time Frame: This outcome will be measured after propofol is administered until the end of the procedure.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Ketamine 0 mg/kg | Ketamine 0.25 mg/kg | Ketamine 0.5 mg/kg | Ketamine 1.0 mg/kg
Number analyzed (Participants) | 14 | 14 | 13 | 14
seconds | 59 (26) | 45 (20) | 57 (19) | 39 (12)

3. Secondary Outcome: Incidence of Adverse Respiratory Events During the Procedure
Description: Any respiratory adverse event including desaturation <95 requiring oxygen administration or need for airway management maneuvers (jaw thrust, bag/mask ventilation) to relieve upper airway obstruction
Time Frame: From induction of anesthesia until endoscopy procedure is complete
Measure: Count of Participants; unit: Participants
Arm/Group | Ketamine 0 mg/kg | Ketamine 0.25 mg/kg | Ketamine 0.5 mg/kg | Ketamine 1.0 mg/kg
Number analyzed (Participants) | 14 | 14 | 13 | 14
Participants
  Desaturation requiring supplemental oxygen | 11 | 10 | 11 | 9
  Need for airway management | 1 | 1 | 2 | 1

4. Secondary Outcome: Incidence of Side Effects and Complications During the Recovery Period
Description: Side effects including:
  hallucinations and/or emergence delirium measured by the Pediatric Anesthesia Emergence Delirium (PAED) scale dizziness nausea and/or vomiting administration of antiemetic pain > 3/10 at any site (measured using age appropriate scale) time to discharge readiness using established criteria reasons for delayed discharge (if any)
Time Frame: From the time procedure is complete until discharge from hospital with an average time of 1 hour.
Measure: Count of Participants; unit: Participants
Arm/Group | Ketamine 0 mg/kg | Ketamine 0.25 mg/kg | Ketamine 0.5 mg/kg | Ketamine 1.0 mg/kg
Number analyzed (Participants) | 14 | 14 | 13 | 14
Participants
  Hallucinations | 0 | 0 | 1 | 0
  Nausea/vomiting | 0 | 0 | 2 | 4
  Dizziness | 6 | 7 | 8 | 9
  Nystagmus/visual disturbance | 3 | 5 | 3 | 9
  Emergence delirium | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From the time patient enters recovery room to discharge from hospital
Arm/Group | Ketamine 0 mg/kg | Ketamine 0.25 mg/kg | Ketamine 0.5 mg/kg | Ketamine 1.0 mg/kg
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/14 | 0/13 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14 | 0/13 | 0/14
Other Adverse Events (participants affected / at risk) | 7/14 | 8/14 | 10/13 | 11/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ketamine 0 mg/kg (N=14) | Ketamine 0.25 mg/kg (N=14) | Ketamine 0.5 mg/kg (N=13) | Ketamine 1.0 mg/kg (N=14)
Hallucinations (Nervous system disorders) | 0 | 0 | 1 | 0
Nausea/vomiting (Gastrointestinal disorders) | 0 | 0 | 2 | 4
Dizziness (Nervous system disorders) | 6 | 7 | 8 | 9
Nystagmus/visual disturbance (Nervous system disorders) | 3 | 5 | 3 | 9
Emergence delirium (Nervous system disorders) | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes